CLINICAL TRIAL: NCT00818116
Title: Visual Function After Implantation of Bilateral AcrySof ReSTOR Aspheric Intraocular Lens (IOL): Postmarket Evaluation
Brief Title: Visual Function Evaluation of Bilateral AcrySof ReSTOR Aspheric IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: China: Ethics Committee, Alcon China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-08-001
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-06

CONDITIONS: Cataracts
Keywords: Cataract; visual acuity; AcrySof ReSTOR Aspheric Intraoculare Lens; Bilateral cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR Aspheric IOL (Experimental): Bilateral implantation with the AcrySof ReSTOR Aspheric Intraocular Lens (IOL)
  Interventions: Device: AcrySof ReSTOR Aspheric IOL

INTERVENTIONS:
Device: AcrySof ReSTOR Aspheric IOL — Bilateral implantation with the AcrySof ReSTOR Aspheric Intraocular Lens (IOL) for the replacement of cataract in the natural lens of the eye.

SUMMARY:
The objective of this study is to evaluate postoperative visual function in patients implanted bilaterally with the ReSTOR Aspheric Intraocular Lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract patients who require natural crystalline lens removal and bilateral Intraocular Lens (IOL) implantation.
* 50~75 years of age
* <1 Diopter of astigmatism preoperatively (before surgery) as measured by Keratometry readings.

Exclusion Criteria:

* Patients with pre-existing conditions that could skew the results.
* Any of conditions before and during surgery specified in the product information.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 eligible patients were enrolled into the study
Pre-assignment Details: Open-label, single arm, non-randomized
Groups:
- ReSTOR Aspheric: Implantation with the AcrySof ReSTOR Aspheric Intraocular Lens (IOL)
Period: Overall Study
Arm/Group | ReSTOR Aspheric
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR Aspheric
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected and Best Corrected Visual Acuities (Near and Distance)
Description: Measurement of uncorrected (without spectacles or other visual corrective devices) and best-corrected (with spectacles or other visual corrective devices)visual acuity at both near and distance. Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 6 Months Following Cataract Surgery
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Aspheric
Number analyzed (Participants) | 34
logMAR
  Near Uncorrected Visual Acuity | 0.02 (0.08)
  Near Best-Corrected Visual Acuity | 0.01 (0.07)
  Distance Uncorrected Visual Acuity | 0.00 (0.07)
  Distance Best-Corrected Visual Acuity | -0.03 (0.07)

ADVERSE EVENTS:
Time Frame: 1 Day, 1 Month, 3 Months, and 6 Months following cataract surgery.
Arm/Group | ReSTOR Aspheric
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReSTOR Aspheric (N=34)
Glare (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No